CLINICAL TRIAL: NCT06348524
Title: Ferumoxytol-enhanced Magnetic Resonance Imaging
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: new IRB not available
Sponsor: Transmed Solutions (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ferumoxytol_2015
Record Dates: First submitted 2023-07-29; First posted 2024-04-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm utilizing ferumoxytol (Experimental)
  Interventions: Drug: Ferumoxytol injection

INTERVENTIONS:
Drug: Ferumoxytol injection — ferumoxytol will assess patency of coronary arteries

SUMMARY:
There are no current alternatives to diagnostic contrast-requiring imaging for patients with an eGFR <30mL/min due to the association of gadolinium-based imaging modalities to nephrogenic systemic fibrosis and iodinated contrast-induced kidney injury. Ferumoxytol-enhanced imaging may offer an alternative approach.

DETAILED DESCRIPTION:
This is a case control study which will assess the resolution by which the coronary arteries can be visualized using ferumoxytol-enhanced cardiac magnetic resonance angiography (fcMRA) in patients with prior regional cardiac ischemia localized by stress-induced echocardiography. Resolution will be compared to invasive coronary arteriography completed in all patients that will be analyzed at the end of the study.

Masked experts will interpret fcMRA images to determine if coronary stenosis is present or absent. By strict definitions, this is a single-arm study. However comparison will be made between fcMRA and invasive coronary arteriography performed in each patient. With a prevalence of disease of approximately 0.35 in the study population, it is anticipated that both sensitivity and specificity of fcMRA to identify the absence of coronary artery stenosis can be calculated.

ELIGIBILITY:
Both female and male participants are being studied aged 18-85 years old with an estimated glomerular filtration rate (eGFR) of less than 30ml/min/1.73 meters squared. Patients will have undergone cardiac screening tests that warrant further evaluation. Patients will be excluded with an eGFR >30ml/min/1.73 meters squared.

Inclusion criteria:

Diagnosis of chronic kidney disease Diagnosis of anemia of chronic kidney disease

Exclusion criteria:

Hypersensitivity to intravenous iron products

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Detect the absence of ≥50% stenosis in the coronary artery tree | 12 months
  This outcome derives from the central hypothesis which states that coronary artery disease can more effectively be excluded in patients with severe chronic kidney disease using ferumoxtyol enhanced cardiac magnetic resonance angiography (fcMRA) rather than non-invasive cardiac testing combined with ICA. The presence or absence of a single 50% stenosis in the region of interest (measured as described above) will be dichotomized (0=absent/ 1= present) from each of the two measures, fcMRA and invasive coronary arteriography

SECONDARY OUTCOMES:
Detect stenosis in proximal and distal segments of the coronary artery tree | 12 months
  The purpose of this secondary outcome is to determine the sensitivity and specificity of fcMRA to detect the absence of lesions exhibiting ≥50% stenosis compared to ICA in proximal and distal arterial segments
Compare ferumoxtyol enhanced magnetic resonance angiography with stress echocardiography | 12 months
  The purpose of this secondary outcome is to determine the sensitivity and specificity of fcMRA to dobutamine stress echocardgiography testing in the assessment of coronary artery stenosis when compared to ICA.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Siedlecki, MD, Principal Investigator — authorized representative

IPD SHARING:
Plan to Share IPD: No